CLINICAL TRIAL: NCT03518476
Title: Evaluation of an Intensive Education Program on the Treatment of Tobacco Use Disorder for Pharmacists: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other); International Islamic University Malaysia (Other); University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Dr. Maguy El Hajj, Associate Professor and Chair of Clinical Pharmacy and Practice Section, Qatar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QatarU
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Pharmacists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in the intervention group will participate in an intensive education program delivered by a multi-disciplinary group of educators, researchers, and clinicians with expertise in tobacco control and tobacco dependence treatment. The program will be delivered over 4 days (run over 2 weekends) with an average of eight contact hours per day (a total of 32 contact hours) at Qatar University.
  Interventions: Behavioral: intensive multi-disciplinary education program on tobacco treatment for pharmacists
- Control arm (Active Comparator): Non-tobacco related training or education sessions will delivered to pharmacists in the control group.
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: intensive multi-disciplinary education program on tobacco treatment for pharmacists — Participants in the intervention group will participate in an intensive education program delivered by a multi-disciplinary group of educators, researchers, and clinicians with expertise in tobacco control and tobacco dependence treatment. The program will be delivered over 4 days (run over 2 weekends) with an average of eight contact hours per day (a total of 32 contact hours) at Qatar University.
  Arms: Intervention arm
Other: Control arm — Participants in control arm will receive a non-tobacco related training or educational session
  Arms: Control arm

SUMMARY:
In Qatar, tobacco use is one of the main causes of premature deaths and preventable diseases. As per the 2013 Global Adult Tobacco Survey (GATS), 12.1% of adults and 20.2% of men in Qatar smoke tobacco, and 55.4% of this smoke an average of 16 cigarettes or more per day. Moreover, 15.7% of school students aged 13 to 15 years currently use some form of tobacco according to the 2013 Global Youth Tobacco Survey (GYTS). In Qatar, tobacco-related diseases including cardiovascular diseases and cancers are highly prevalent. In an effort to reduce tobacco use, Qatar has ratified the WHO Framework Convention on Tobacco Control (FCTC) and has implemented many tobacco control initiatives. In spite of these measures, tobacco use is still rising in Qatar. Pharmacists practicing in retail/community pharmacy are often the first port of call for individuals requiring health advice in general. Evidence has proven that they have a pivotal role in health promotion and disease prevention including tobacco cessation. Hence, pharmacists have excellent opportunities to reduce tobacco use in Qatar. Yet, ambulatory and community pharmacists in Qatar are not sufficiently contributing to tobacco control. Based on published data, only 21% of community pharmacists in Qatar always or most of the time ask patients about their smoking status. Furthermore, when asked about their smoking cessation training, 89% of pharmacists did not receive any kind of education or training about smoking cessation counseling in the past. In an effort to build the capacity of pharmacists in Qatar, the aim of the proposed study is to design, implement and evaluate an intensive education program on tobacco treatment for pharmacists in Qatar. The study will be a prospective randomized controlled trial comparing the effectiveness of the education program on pharmacists' tobacco cessation-related knowledge, attitudes, self-efficacy, and skills.

ELIGIBILITY:
Inclusion Criteria:

* Retail/community pharmacists practicing in Qatar will be eligible for participation in the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
tobacco related knowledge post program | at the end of the program (+ 1 DAY POST THE PROGRAM)
  This outcome will be assessed using a survey instrument
tobacco cessation related skills difference between the 2 groups | at the end of the program (+ 1 DAY AFTER THE PROGRAM)
  This outcome will be assessed using OSCE (Objective Structured Clinical Examination).
  Pharmacist's practical skills in the delivery of effective tobacco cessation will be assessed through the use of a performance-based assessment such as Objective Structured Clinical Examination (OSCE). Examples of skills to be assessed include communication skills in general, counselling skills, law and professional ethics, and interviewing skills. We propose a 5 to 8 station OSCE that will target core competencies and skills covered in the program. In the OSCE, each participant will be allocated 10 mins to interact with a standardized patient who will be trained using a validated script. Performance of participants will be assessed using validated assessment checklists.

SECONDARY OUTCOMES:
tobacco cessation related skills difference between the 2 groups | 3-6 months post intervention
  The secondary endpoint of the study will be the performance difference in relation to skills in the practice setting between the intervention and the control groups assessed using the simulated client approach.
  In this phase, the study will evaluate whether participants in intervention and control groups will offer appropriate tobacco cessation counseling and will recommend proper tobacco cessation aids in their practice setting. Using a simulated client approach to data collection 3 to 6 months post program, the study will assess the quality of advice and recommendations of participants given to simulated clients asking for help in quitting smoking. Simulated clients using designed and validated case scenarios will visit participants in both groups. The clients will be selected to resemble the sociodemographic and practice characteristics of Qatar population and residents. Objective assessment forms will be developed using tobacco cessation guideline
tobacco related self-efficacy difference between the 2 groups | at the end of the program (+ 1 DAY POST THE PROGRAM)
  This outcome will be assessed using a survey instrument
tobacco related attitudes difference between the 2 groups | at the end of the program (+ 1 DAY POST THE PROGRAM)
  This outcome will be assessed using a survey instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Qatar Univeristy, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Hajj MS, Awaisu A, Nik Mohamed MH, Saleh RA, Al Hamad NM, Kheir N, Mahfoud ZR. Assessment of an intensive education program for pharmacists on treatment of tobacco use disorder using an objective structured clinical examination: a randomized controlled trial. BMC Med Educ. 2022 Apr 18;22(1):289. doi: 10.1186/s12909-022-03331-9. PMID 35436957
- [Derived] El Hajj MS, Awaisu A, Kheir N, Mohamed MHN, Haddad RS, Saleh RA, Alhamad NM, Almulla AM, Mahfoud ZR. Evaluation of an intensive education program on the treatment of tobacco-use disorder for pharmacists: a study protocol for a randomized controlled trial. Trials. 2019 Jan 8;20(1):25. doi: 10.1186/s13063-018-3068-7. PMID 30621772